CLINICAL TRIAL: NCT00228371
Title: Assessment of Subthalamic Nucleus Stimulation in Drug Resistant Epilepsy Associated With Dopaminergic Metabolism Deficit. A Randomized, Double Blind, Controlled Trial.
Brief Title: STIMEP : Assessment of Subthalamic Nucleus Stimulation in Drug Resistant Epilepsy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: insufficent enrolement
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DCIC 03 23
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Epilepsy; Drug Resistant
Keywords: Epilepsy; deep brain stimulation; Subthalamic nucleus; Drug resistant epilepsy
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): The stimulator is switch ON during the first phase of the cross-over and switch OFF during the second phase
  Interventions: Device: Neurostimulation
- 2 (Other): The stimulator is switch OFF during the first phase of the cross-over and switch ON during the second phase
  Interventions: Device: Neurostimulation

INTERVENTIONS:
Device: Neurostimulation — High frequency neurostimulation of subthalamic nucleus : quadrupolar electrode, type 3389, n° : I7 02 08 39709 158, Medtronic, Minneapolis, USA
  Other Names: Neurostimulation of subthalamic nucleus

SUMMARY:
The aim of this study is to evaluate the effectiveness and the safety of deep brain stimulation in drug resistant epilepsy.

This is a double blind, controlled and randomized clinical trial with two cross-over groups and four phases.

Phase 1 : base line, open phase consisting of follow-up of patients with their standard treatment.

Phase 2 : Randomisation, lead implantation, followed by 3 months wash out period with the stimulator switch OFF.

Phase 3 : cross-over, double blind phase : 3 months with stimulator switch ON or OFF depending on randomization allocation, followed by 3 months with the stimulator switch on the opposite position. The placebo consisting of turn OFF the stimulator.

Phase 4 : open phase, one year follow-up of all patients with the stimulator switch ON.

DETAILED DESCRIPTION:
The experimental work performed for more than 15 years by several research teams shows in animal models of epilepsy, that several circuits of basal ganglia are involved in the control of epilepsy seizures. The existence of those circuits leads to the possibility of therapeutic applications in particular deep brain stimulation.

Preliminary results (Benabid et al, 2002) (Chabardes et al , 2002) suggest that the neuromodulation of basal ganglia and in particular the subthalamic nucleus and the substantia nigra pars reticulata could have a therapeutic effects in patients with drug resistant epilepsy and no possibility of resection surgery.

This is a double blind, controlled and randomized clinical trial with two cross-over groups and four phases.

Phase 1 : base line, open phase consisting of follow-up of patients with their standard treatment.

Phase 2 : Randomisation, lead implantation, followed by 3 months wash out period with the stimulator switch OFF.

Phase 3 : cross-over, double blind phase : 3 months with stimulator switch ON or OFF depending on randomization allocation, followed by 3 months with the stimulator switch on the opposite position.

Phase 4 : open phase, one year follow-up of all patients with the stimulator switch ON.

There are two differents groups at phase 3 :

* Group A : 10 patients with the stimulator switch ON for three months and switch OFF for the next three months.
* Group B : 10 patients with the opposite sequence, OFF and ON.

Main objective :

- To show that high frequency deep brain stimulation of the subthalamic nucleus decrease the frequency of epileptic seizure compared with no stimulation.

Secondary objectives :

* To show that high frequency deep brain stimulation of the subthalamic nucleus improve the quality of life.
* To describe the side effects of this device and compare with those described in Parkinson patients. In particular to check the onset of dyskinesia related to dopamine.
* To compare the distribution of seizure frequency after stimulation to the base line.
* To show that the number of patients responding to treatment are higher in the group with stimulator switch ON than in the group with the stimulator turn OFF.
* To compare the number of days without seizure with the stimulator switch ON or OFF.
* To evaluated the neuropsychologic effect induced by the neurostimulation
* To quantify the types and the ratio of different seizures during the ON phase and the OFF phase.
* To monitor the secondary drug use during the study.

Control visits : all patients will have a control visit every 4 weeks during the study.

ELIGIBILITY:
Inclusion Criteria:

* Epilepsy resistant to antiepileptic drug and dopaminergic D2 agonist.
* No curative exeresis surgery possible
* Metabolism deficiency of DOPA above 1 DS, evaluated by Positron Emission Tomography (PET) using fluorodopa
* Age ranging from 18 to 50
* capacity to consent
* Affiliation to the French Social Security

Exclusion Criteria:

* pregnant woman or nursing mother
* change of antiepileptic, 30 days before base line
* convulsive "etat de mal" that requires an hospitalisation, 30 days before base line

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
- Daily seizure frequency at each phase | at each phase

SECONDARY OUTCOMES:
The number of days without seizure during each phase | at each phase
Quality of life : SEALS, QOLIE-31 and NHP scales | at each phase
Neuropsychological test : WAIS, GROBER and Busckhe, Wisconsin Card Sorting Test, TRAIL test, LURIA test, Beck Depression Inventory, verbal flow test, empathy test | at each phase

CONTACTS AND LOCATIONS:
Overall Officials: Stephan CHABARDES, Dr, Principal Investigator — University Hospital of Grenoble, Neuro surgery
Locations (3):
- France (3):
  - University Hospital of Grenoble, Grenoble, Isere
  - University Hospital of Rennes, Rennes
  - University Hospital of Strasbourg, Strasbourg

REFERENCES:
- [Background] Alexander GE, Crutcher MD. Functional architecture of basal ganglia circuits: neural substrates of parallel processing. Trends Neurosci. 1990 Jul;13(7):266-71. doi: 10.1016/0166-2236(90)90107-l. PMID 1695401
- [Background] Ardouin C, Pillon B, Peiffer E, Bejjani P, Limousin P, Damier P, Arnulf I, Benabid AL, Agid Y, Pollak P. Bilateral subthalamic or pallidal stimulation for Parkinson's disease affects neither memory nor executive functions: a consecutive series of 62 patients. Ann Neurol. 1999 Aug;46(2):217-23. doi: 10.1002/1531-8249(199908)46:23.0.co;2-z. PMID 10443887
- [Background] Benabid AL, Koudsie A, Benazzouz A, Vercueil L, Fraix V, Chabardes S, Lebas JF, Pollak P. Deep brain stimulation of the corpus luysi (subthalamic nucleus) and other targets in Parkinson's disease. Extension to new indications such as dystonia and epilepsy. J Neurol. 2001 Sep;248 Suppl 3:III37-47. doi: 10.1007/pl00007825. PMID 11697687
- [Background] Benabid AL, Minotti L, Koudsie A, de Saint Martin A, Hirsch E. Antiepileptic effect of high-frequency stimulation of the subthalamic nucleus (corpus luysi) in a case of medically intractable epilepsy caused by focal dysplasia: a 30-month follow-up: technical case report. Neurosurgery. 2002 Jun;50(6):1385-91; discussion 1391-2. doi: 10.1097/00006123-200206000-00037. PMID 12015863
- [Background] Chabardes S, Kahane P, Minotti L, Koudsie A, Hirsch E, Benabid AL. Deep brain stimulation in epilepsy with particular reference to the subthalamic nucleus. Epileptic Disord. 2002 Dec;4 Suppl 3:S83-93. PMID 12495878
- [Background] Chkhenkeli SA, Chkhenkeli IS. Effects of therapeutic stimulation of nucleus caudatus on epileptic electrical activity of brain in patients with intractable epilepsy. Stereotact Funct Neurosurg. 1997;69(1-4 Pt 2):221-4. doi: 10.1159/000099878. PMID 9711758
- [Background] Cooper IS, Amin I, Gilman S. The effect of chronic cerebellar stimulation upon epilepsy in man. Trans Am Neurol Assoc. 1973;98:192-6. No abstract available. PMID 4206369
- [Background] DeLong MR. Primate models of movement disorders of basal ganglia origin. Trends Neurosci. 1990 Jul;13(7):281-5. doi: 10.1016/0166-2236(90)90110-v. PMID 1695404
- [Background] Dematteis M, Kahane P, Vercueil L, Depaulis A. MRI evidence for the involvement of basal ganglia in epileptic seizures: an hypothesis. Epileptic Disord. 2003 Sep;5(3):161-4. PMID 14684352